CLINICAL TRIAL: NCT05494528
Title: An, Open-label, Multicenter, Randomized, Active Control Study, Comparing P1101 Monotherapy to Entecavir Monotherapy in Patients With HBeAg-negative Chronic Hepatitis B Under Long-term Nucleos(t)Ide Analogue Therapy
Brief Title: Comparing P1101 to Entecavir in Patients With HBeAg(-) Hepatitis B Under Long-term Nucleos(t)Ide Analogue Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202003098MIPD; A18-I02 (Other: PharmaEssentia Corporation)
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-03

CONDITIONS: Chronic Hepatitis B Virus Infection
Keywords: Ropeginterferon alpha-2b; Hepatitis B; Entecavir; HBeAg-negative; Nucleoside Analogue Therapy
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropeginterferon alfa-2b monotherapy (Experimental): Subjects will be treated with 450 µg of Ropeginterferon alfa-2b every two weeks
  Interventions: Drug: Ropeginterferon alfa-2b
- Entecavir monotherapy (Active Comparator): Subjects will be treated with 0.5 mg of Entecavir monotherapy once per day
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Ropeginterferon alfa-2b — Ropeginterferon alfa-2b 450 µg subcutaneous injection every two weeks
  Other Names: P1101
  Arms: Ropeginterferon alfa-2b monotherapy
Drug: Entecavir — Entecavir 0.5 mg once per day
  Arms: Entecavir monotherapy

SUMMARY:
This is an open-label, multicenter, randomized, active control study, comparing P1101 monotherapy to entecavir monotherapy in patients with HBeAg-negative chronic hepatitis B under long-term nucleos(t)ide analogue therapy.

DETAILED DESCRIPTION:
Eligible patients will be randomized in a 2:1 ratio (P1101 monotherapy vs. Entecavir monotherapy) using a computer-generated permuted block randomization scheme.

Subjects will be treated with 450 µg of P1101 every two weeks or with 0.5 mg of Entecavir monotherapy once per day. Primary endpoint will be evaluated at week 48. Subjects will receive treatment with a total duration of 72 weeks. The follow-up (treatment-free) period is 24 weeks following completion of treatment. Switch from the other nucleos(t)ide analogue therapy to entecavir will occur at week 0 (Randomization), while the dose of Entecavir will be 0.5 mg.

ELIGIBILITY:
Inclusion Criteria:

* Adults with age 20-75 years old; Subjects who are over 70 years of age must be in generally good health;
* Confirmed diagnosis of chronic hepatitis B (CHB) virus infection: with positive HBsAg ≧ 6 months prior to the study entry;
* Quantitative HBsAg level < 1,500 IU/ml at screening;
* Confirmed HBeAg (-) at screening;
* Stable disease: ALT < 3 x upper limit of normal (ULN), total bilirubin < 1.5 × ULN (except in Gilbert syndrome) and direct bilirubin < ULN at screening, serum HBV DNA < 50 IU/mL for ≧ 1 year prior to study entry;
* Stable treatment with nucleos(t)ide regimen (adefovir, entecavir, tenofovir or one of the following combinations: entecavir/adefovir or entecavir/tenofovir) for at least 2 years prior to study entry;
* Interferon treatment naïve;
* Normal fundoscopic examination by ophthalmologist at screening; defined as no significant or major fundoscopic findings including but not limited to retinal exudates, hemorrhage, detachment, neovascularization, papilloedema, optic atrophy, microaneurysms and macular changes;
* Be able to attend all scheduled visits and to comply with all study procedures;
* Be able to provide written informed consent.

Exclusion Criteria:

* HBeAg-positive chronic hepatitis B;
* Documented history of drug resistance to any nucleoside/ nucleotide analogue;
* History of treatment with lamivudine or telbivudine prior to the study entry;
* Clinically significant abnormalities, other than HBV infection, based upon the results of a medical history, physical examination, vital signs, and a 12-lead electrocardiogram (ECG) at screening as determined by the investigator;
* Other form of significant chronic liver disease apart from chronic hepatitis B infection; Severe steatohepatitis by ultrasound or other examinations at the discretion of investigators;
* Liver cirrhosis;
* Known positive for anti-HIV;
* Positive for anti-hepatitis C virus(HCV), Subject could be enrolled if no HCV RNA detected within 1 year；
* Co-infection with hepatitis D;
* One of clinically significant abnormal laboratory test result at screening: white blood cell (WBC) < 3,000/mm^3, absolute neutrophil count (ANC) < 1500/mm^3, Hgb < 10g/dL, platelet < 90,000/mm^3, estimated Glomerular filtration rate < 60 mL/min;
* History of significant alcohol or illicit drug abuse within six months prior to the screening visit (alcohol consumption of more than fourteen units of alcohol per week [1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]) or refusal to abstain from illicit drugs and minimize alcohol consumption throughout the study;
* History of severe allergic or hypersensitivity reactions (e.g bronchospasm, angioedema), asthma, or anaphylaxis
* Therapy with any systemic anti-viral treatment (except for treatment for HBV), anti-neoplastic, immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) and immunosuppressants within 1 month (3 months for those with long elimination half-lives) prior to the first dose of study drug;
* Use of an investigational drug within the last 4 weeks;
* Any history or presence of poorly controlled or clinically significant medical conditions that are not suitable to receive interferon-based treatment, at the discretion of the investigator: major psychiatric (including but not limited to those with severe depression, severe bipolar disorder, schizophrenia, suicidal ideation or history of suicidal attempt),neurological, cardiovascular (e.g. uncontrolled hypertension), pulmonary (including but not limited to chronic obstructive lung disease), hematological, immunologic, endocrine, metabolic (e.g. diabetes mellitus with HbA1C > 8.0%), autoimmune disease, thyroid or other uncontrolled systemic disease, coagulation disorders or blood dyscrasias;
* A depot injection or an implant of any drug within 3 months prior to administration of study medication, other than contraception or hyaluronic acid injections in joints for osteoarthritis;
* History of solid organ transplantation;
* History of malignancy diagnosed or treated within 5 years prior to screening (except for recent localized treatment of squamous or noninvasive basal cell skin cancers; cervical carcinoma in situ), cancer survivors not on maintenance therapy within the past 5 years;
* History of opportunistic infection (e.g., invasive candidiasis or pneumocystis pneumonia)
* Serious localized infection (e.g., cellulitis, abscess) or systemic and life-threatening infection (e.g., septicemia) within the 3 months prior to screening;
* Pregnant subjects. Female subjects or the spouse of male subjects, with child-bearing potential who are unwilling or unable to practice adequate contraception, defined as vasectomy in men, tubal ligation in women, or use of condoms and spermicides, or birth control pills, or intrauterine devices from 4 weeks prior to Day 1 until 90 days after the last dose of study drug.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Undetectable HBsAg | Week 48
  HBsAg loss at week 48

SECONDARY OUTCOMES:
Undetectable HBsAg | weeks 72 and 96
  HBsAg loss at weeks 72 and 96
HBsAg level | weeks 12, 24, 48, 72 and 96
  HBsAg reduction > 1 log from baseline to weeks 12, 24, 48, 72 and 96
HBsAg and anti-HBs level | weeks 48, 72 and 96
  HBsAg seroconversion at weeks 48, 72 and 96
HBsAg level | weeks 12, 24, 48, 72, and 96
  Mean HBsAg decline from baseline to weeks 12, 24, 48, 72, and 96
Reappearance of HBsAg | weeks 72 and 96
  HBsAg seroreversion at weeks 72 and 96
HBV DNA level | week 96
  Percentage of subjects with HBV DNA > 2,000 IU/ml at week 96
HBV DNA and alanine aminotransferase (ALT) level | week 96
  Percentage of subjects with HBV DNA > 2,000 IU/ml and ALT > 2x ULN at week 96
Sustained suppression of HBV DNA | week 96
  Sustained suppression of HBV DNA less than the lower limit of qualification at week 96.
HBeAg level | weeks 72 and 96
  To compare the proportion of HBeAg seroreversion and seroconversion at weeks 72 and 96 across treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Jen Liu, Principal Investigator — National Taiwan University Hospital
Locations (5):
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No